CLINICAL TRIAL: NCT01424904
Title: DGB-01 Effects on Endurance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Black (Other)
Collaborators: Immunotec Inc. (Industry)
Responsible Party: Sponsor-Investigator, William Black, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11-0626-F1V
Record Dates: First submitted 2011-08-19; First posted 2011-08-29 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Fatigue
Keywords: Ergogenic aid; Exercise endurance; High performance; Time trial performance; Glutathione
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- DGB-01 (Experimental): All subjects will receive DGB-01 during the study. Approximately one-half of the subjects during the first period and the other half during the second period.
  Interventions: Dietary Supplement: DGB-01 Supplementation

INTERVENTIONS:
Dietary Supplement: DGB-01 Supplementation — Approximately one-half of the subjects will initially receive DGB-01. The other half of the subjects will receive casein. Investigators and subjects are blinded to the product the subject is receiving. Subjects will be asked to consume one pouch of their assigned study product twice daily for four weeks.
  Subsequently, all subjects will undergo a supplement-free washout period of at least four weeks duration. Following the washout period, the subjects who originally received DGB-01 will receive casein and the subjects who originally received casein will receive DGB-01. Subjects will be asked to consume one pouch of their assigned study product twice daily for four weeks.

SUMMARY:
The purpose of this research is to evaluate the effects of DGB-01 on performance of a 40-km time trial in trained male cyclists. The investigators believe that DGB-01 will improve performance on the time trial as measured by a reduction in the amount of time required to complete the distance, using a computerized cycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males who are trained cyclists with a maximal oxygen uptake relative to body weight equal to or greater than 45 ml O2/kg/min.
* Subjects must be in the competitive phase of their annual training cycle.
* Between ages of 18-60
* Availability- commitment of the subject/expected participation in the study for 97 days.

Exclusion Criteria:

* Specific allergy to milk proteins (this is different from lactose intolerance)
* Use of immunosuppressive medication in the case of organ transplants
* Planned surgeries.
* Kidney disorders
* Use of antihypertensive medications
* Cardiovascular disease
* Abnormal BUN, creatinine, hemoglobin, or hematocrit
* Body weight greater than 285 pounds
* A protein-restricted diet
* Subjects currently using dry whey protein supplements, N-acetylcysteine, or alpha-lipoic acid supplements. The wash-out period is 1 month for any of these supplements.
* All medications that can interfere with muscle mass such as corticosteroids (e.g. prednisone), testosterone replacement or anabolic drugs such as Megace

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The efficacy of DGB-01 in promoting exercise endurance will be measured by cycling performance on a standardized 40-km time trial course. | Individual participants will be followed for the duration of study enrollment, an expected average of 97 days. The study will remain open for up to 2 years or until subject number requirement is met.
  Time to complete the 40km time trial for subjects with DGB-01 intervention in period 1 (minimum 4 weeks of supplementation) versus the time for time trial completion of these subjects with casein in period 2 (minimum of 4 weeks of supplementation); Between the two periods with supplementation, there will be a washout period of a minimum 4 weeks; Results of time trial for subjects with DGB-01 intervention in period 2 (minimum 4 weeks of supplementation) versus the time trial completion of these subjects with casein in period 1 (minimum 4 weeks supplementation).

SECONDARY OUTCOMES:
Change in markers of plasma thiol status over the course of each time trial | Individual participants will be followed for the duration of study enrollment, an expected average of 97 days. The study will remain open for up to 2 years or until subject number requirement is met.
  * A) Plasma samples will be obtained before and during the final minute of each time trial. These samples will be stored at -80oC for no longer than 14 days to prevent sample deterioration.
  * B) All samples will be analyzed for glutathione (GSH), oxidized glutathione (GSSG), cysteine (CySH), cystine (CySS), and cysteine-glutathione disulfide (CySSG) using high-performance liquid chromatography (Clinical Biomarkers Laboratory, Emory University, Atlanta, GA). Total glutathione (TGSH) will be calculated as GSH + 2•GSSG + CySSG. Total cysteine (TCyS) will be calculated as CySH + 2•CySS + CySSG.
Outcome from specific questionnaires | Individual participants will be followed for the duration of study enrollment, an expected average of 97 days. The study will remain open for up to 2 years or until subject number requirement is met.
  A) The Standardized Overtraining Questionnaire of The French Society for Sports Medicine (SFMS) B) Foster's Psychological Complaint Index C) Classification of Muscle Soreness

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reid, Ph.D, Principal Investigator — University of Kentucky, Dept of Physiology; William Black, MD, Principal Investigator — University of Kentucky, Dept of Physiology
Locations (1):
- Center for Clinical and Translational Science, Lexington, Kentucky, United States